CLINICAL TRIAL: NCT04168905
Title: Multi-Center, Prospective, Randomized,Controlled Trial to Evaluate the Efficacy of Cyclical Topical Wound Oxygen Therapy (TWO2) in the Treatment of Chronic Wounds
Brief Title: Cyclical Topical Wound Oxygen Therapy (TWO2) in the Treatment of Chronic Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Lishui Central Hospital，Lishui Hospital of Zhejiang University (Unknown); Ningbo No.6 Hospita (Unknown); Inner Mongolia People's Hospital (Other); Qingdao Hiser Hospital Affiliated to Qingdao University (Unknown); No.1 Hospital of Honghezhou (Unknown); Pingdingshan City Hospital of Traditional Chinese Medicine (Unknown); The department of burns of the first affiliated hospital of SUN YAT-Sen university (Unknown); Hangzhou Enhua Hospital (Unknown); The 1st affiliated hospital of Jinzhou Medicine University (Unknown); Suzhou Municipal Hospital (Other); Suzhou Science and Technology City Hospital (Unknown); Shanghai Deji Hospital (Unknown); Wujin people hospital of Changzhou city (Unknown); Affiliated hospital of Xinyang vocational technical institute (Unknown); Sichuan Provincial People's Hospital (Other); uncheng Central Hospital of Shanxi Province (Unknown); The Second Affiliated Hospital of Dalian Medical University (Other); First Affiliated Hospital of Jinan University (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-236
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-05

CONDITIONS: Evaluate the Efficacy of Cyclical Topical Wound Oxygen Therapy in the Treatment of Chronic Wounds
Keywords: chronic wounds; Topical wound oxygen therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): After receiving standard treatment and AOTI Inc. TWO2 topical oxygen therapy equipment training, patients will apply themselves oxygen therapy at home for 5 days a week, 90 minutes a day, rest for 2 days, and follow-up once a week. A total of 12 weeks of treatment, or recieving treatment till wound healed.
  Interventions: Device: AOTI Inc. TWO2 topical oxygen therapy equipment
- Controlled arm (Placebo Comparator): patients receive standard treatment.
  Interventions: Device: AOTI Inc. TWO2 topical oxygen therapy equipment

INTERVENTIONS:
Device: AOTI Inc. TWO2 topical oxygen therapy equipment — Patients will apply themselves oxygen therapy at home for 5 days a week, 90 minutes a day, rest for 2 days, and follow-up once a week. A total of 12 weeks of treatment, or recieving treatment till wound healed.

SUMMARY:
To evaluate the efficacy and clinical satisfaction of topical oxygen therapy (LOT) in chronic wounds (including patients and medical staff), and explore its possible mechanism.

DETAILED DESCRIPTION:
A multi-center open randomized controlled study was conducted. A total of 240 subjects were expected to be accepted. Patients receiving normative wound treatment received cyclic topical oxygen therapy, not excluding the treatment of other diseases.

After signing the informed consent, the patients were randomly divided into the treatment group and the control group. The total treatment time was 12 weeks or the wound healed completely. The enrollment examination included lower limb arteriovenous examination (including B-mode ultrasound, ankle-brachial index), and other related necessary examinations (such as biopsy excluding malignant tumors; blood routine, bacterial culture excluding wound infection; vibration area detection excludes peripheral neuropathy). Relevant examinations and records were made at each time point, including pre-admission and weekly follow-up days. Wound area measurement, image data collection, wound analysis, secretion detection, patient pain score and satisfaction survey, medical staff evaluation were required at each time point. Every patient in the group and the follow-up day should be treated according to the guidance of the doctor according to the type of wound, including wet wound treatment, debridement, decompression, stress treatment and so on.

ELIGIBILITY:
Inclusion Criteria:

①18 years old or older, regardless of gender;

②It was clinically diagnosed as chronic lower limb wound, which was located below the thigh.

Patients who received mainly etiological treatment, wet dressing change and necessary decompression for more than 2 weeks had no obvious wound healing tendency;

③Understanding the experimental conditions, Patients are willing to participate in and cooperate with the experimental treatment, and sign the informed consent.

Exclusion Criteria:

1. Edema of lower extremity caused by cardiac insufficiency;
2. patients with venous thrombosis of lower extremity;
3. Diabetics with poor blood glucose control: FBS>=8mmol/L; Blood glucose 2h after meal>=10.0mmol/L; HbA1c >= 9%
4. Participated in similar clinical trials in the last three months; Patients with lower extremity arterial occlusion requiring lower extremity vascular surgery;
5. Patients with wound infection requiring systemic antibiotic therapy;
6. Dry scab or necrotic tissue covered more than 50% of the wound, and was not suitable or refused to accept debridement treatment.
7. Immunodeficiency patients
8. Patients with malignant change of wound or with malignant lesions
9. Patients with wound area greater than 10 cm*10 cm;
10. the wound is deep into sclerotin,articular cavity and body cavity;
11. The wound with sinus tract;
12. patients with serious hepatic dysfunction and malnutrition;
13. Patients with mental or other problems and unable to self-manage equipment
14. Treatment of patients with poor compliance.
15. The researchers think there are other reasons which the patients cannot participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Wound healing area | once a week
  The area of wound healing and the appearance of the wound were observed and recorded with each dressing change, and the pictures were collected.
Wound healing rate | once a week
  Percentage of wound healing, percentage of wound healing at each time point were recorded, and the calculation of wound area was evaluated by measuring tools issued by bidders.
Wound healing time | Under 12 weeks
  Record of 100% healing wound

CONTACTS AND LOCATIONS:
Overall Officials: Han Chunmao, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affilated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
We will share our study protocol and results without the patients' privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After our paper's publication.

REFERENCES:
- [Result] Frykberg RG, Franks PJ, Edmonds M, Brantley JN, Teot L, Wild T, Garoufalis MG, Lee AM, Thompson JA, Reach G, Dove CR, Lachgar K, Grotemeyer D, Renton SC; TWO2 Study Group. A Multinational, Multicenter, Randomized, Double-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy of Cyclical Topical Wound Oxygen (TWO2) Therapy in the Treatment of Chronic Diabetic Foot Ulcers: The TWO2 Study. Diabetes Care. 2020 Mar;43(3):616-624. doi: 10.2337/dc19-0476. Epub 2019 Oct 16. PMID 31619393